CLINICAL TRIAL: NCT07298096
Title: A Prospective Single Center, Single Arm, Single-institution Registry That Aims to Assess the Safety and Quality of Life Benefits of Computer-assisted Vacuum Thrombectomy (CAVT) in the Treatment of Cancer Patients With Intermediate Risk Pulmonary Embolism (PE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0830; NCI-2025-08931 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Penumbra Element Sheath (Experimental)
  Interventions: Procedure: Aspiration Thrombectomy

INTERVENTIONS:
Procedure: Aspiration Thrombectomy — All participants in this study will undergo standard of care aspiration thrombectomy.

SUMMARY:
The goal of this clinical research study is to gather information about the quality of life benefits of cancer patients with intermediate risk PE who underwent thrombectomy. The safety of thrombectomy in this patient population will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

To assess the change in the Post Venous Thromboembolism Functional Status (PFVS, see Appendix) score at the time of discharge.

Secondary Objectives:

1. To evaluate quality of life outcomes in patients undergoing thrombectomy by assessing changes in RV/LV ratio from baseline to 48 hours and 90 days post-procedure.
2. To compare PE-related mortality versus all-cause mortality.
3. To assess the incidence of device-related complications and rate of major bleeding events.
4. To assess safety by determining the incidence of major adverse events within 7 days post-treatment.
5. To compare pre- and post-procedure oxygen requirements and six-minute walk test (6MWT) performance in ambulatory patients.
6. To evaluate radiographic changes over time on CT imaging, including parenchymal perfusion and RV/LV ratio in patients undergoing different treatment, at three-time points baseline, 48 hours, and 90 days.
7. To compare BORG Dyspnea Scale scores between pre- and 90-day post-treatment.
8. To evaluate the rate of PE recurrence within 90 days.
9. To evaluate changes in residual volume of PE from baseline to follow-up imaging.
10. To assess the incidence and severity of bleeding events using the BARC (Bleeding Academic Research Consortium) classification, and to explore associations between bleeding events and patients' chemotherapy or immunotherapy regimens through subgroup analysis.
11. To characterize the histopathologic features of retrieved thrombus specimens, categorizing them as either bland thrombus or tumor thrombus, and further classifying tumor thrombi by histologic origin, such as gastrointestinal (GI) or genitourinary (GU) malignancies.
12. To evaluate the reduction in RV/LV ratio on 48-hour post-treatment CT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with current or prior diagnosis of cancer
2. Confirmed PE, based on computed tomographic pulmonary angiography (CTPA) imaging showing a filling defect in at least one main or proximal lobar pulmonary artery
3. Classification of intermediate risk PE as defined by the institutional PERT algorithm
4. Candidate for standard of care pulmonary thrombectomy
5. Age greater than or equal to 18 years. The devices for mechanical thrombectomy are not suitably sized for pediatric patients.
6. ECOG performance status less than or equal to 3
7. Patients must have adequate organ and marrow function as defined below:

   1. absolute neutrophil count ≥ 1,000/mcL
   2. Platelets ≥ 30,000/mcL
8. As these procedures can be performed without the use of iodinated contrast, there are no specific requirements for renal function
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization. Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization.
10. All lines of prior systemic therapy are permissible. Standard concurrent chemotherapy, immunotherapy, or targeted therapy are permissible.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Hemodynamic instability with any of the following present:

   1. Cardiac arrest
   2. Obstructive shock or persistent hypotension defined as systolic blood pressure (BP) <90 mmHg or an acute drop in systolic BP ≥40 mmHg for >15 min, or requiring vasopressor or inotropic support to achieve a systolic BP ≥90 mmHg
2. Patients on ECMO
3. History, imaging or hemodynamic findings consistent with chronic thromboembolic pulmonary hypertension (CTEPH) or chronic thromboembolic disease (CTED) diagnosis
4. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, that catheter-based intervention is not appropriate for the patient

   a. Including but not limited to large volume lung metastases, especially in vascular distribution, large volume pulmonary infarct
5. Allergy, hypersensitivity, or heparin induced thrombocytopenia (HIT)
6. Severe active infection (e.g. sepsis) requiring treatment at time of enrollment
7. Absolute neutrophil count <1000 mm3 within 6 weeks of screening
8. Life expectancy <90 days
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Varshana Gurusamy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org